CLINICAL TRIAL: NCT02323724
Title: APPLICATION OF MOLECULAR TECHNIQUES FOR IMPROVING THE DIAGNOSIS AND TREATMENT OF NODULAR THYROID LESIONS.
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Rosa Bella Cueto, Coordinator of Pathology, Corporacion Parc Tauli
Other Study IDs: 2014/617
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Papillary Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Selected Papillary carcinoma: Cases with histological diagnosis of papillary carcinoma (CP) and previous cytological diagnosis in groups III, IV and V Bethesda, collected between October 1989 and July 2014 in Corporació Parc Taulí.
  Interventions: Genetic: BRAF V600E mutation by pyrosequencing technique

INTERVENTIONS:
Genetic: BRAF V600E mutation by pyrosequencing technique

SUMMARY:
To determine the improvement in diagnosis of papillary carcinoma by detecting mutation V600E BRAF in retrospective cases with inconclusive cytologic diagnosis (categories III, IV and V of Bethesda System)

DETAILED DESCRIPTION:
Aim of the study To determine the improvement in diagnosis of papillary carcinoma by detecting mutation V600E BRAF in retrospective cases with inconclusive cytologic diagnosis (categories III, IV and V of Bethesda System).

Design: Retrospective observational study. Scope: The study will be peformed at the Pathology Service, from cytological samples and paraffin file post-diagnosis. Mutations are detected by pyrosequencing technique.

Subject of study:

Cases with histological diagnosis of papillary carcinoma (CP) and previous cytological diagnosis in groups III, IV and V Bethesda, collected between October 1989 and July 2014 in Corporació Parc Taulí.

Methodology:

* Identification of cases
* Detection of BRAF V600E mutation, initially in histological material from the surgical specimen, and if present, detection in cytological material.

The statistical analysis will use SPSS. Univariate and bivariate analysis will be done. Results will be presented in the form of frequency tables and percentages for qualitative variables and by average, median and standard deviation for quantitative variables. Pearson chi-square or Fisher's exact test will be applied. The Student t test or the Mann-Whitney test will be performed for quantitative variables.

ELIGIBILITY:
Inclusion Criteria:

* Cases with histological diagnosis of papillary carcinoma (CP) and previous cytological diagnosis in groups III, IV and V Bethesda, collected between October 1989 and July 2014 in Corporació Parc Taulí

Exclusion Criteria:

* Non available cytological or histological material

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases with histological diagnosis of papillary carcinoma (CP) and previous cytological diagnosis in groups III, IV and V Bethesda, collected between October 1989 and July 2014 in Corporació Parc Taulí
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Improvement in diagnosis | 6 months
  To determine the improvement in diagnosis of papillary carcinoma by detecting mutation V600E BRAF in retrospective cases with inconclusive cytologic diagnosis (categories III, IV and V of Bethesda System).

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain